CLINICAL TRIAL: NCT04064177
Title: Non-invasive Continuous Cardiac Output Monitoring in Preterm Infants Study
Acronym: NICCOM
Status: Recruiting | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19QC5170
Record Dates: First submitted 2019-08-06; First posted 2019-08-21 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Output, Low; Cardiac Output, High; Blood Pressure
Keywords: Blood Pressure
MeSH Terms: conditions — Cardiac Output, Low; Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Babies (24-42 weeks): All babies born between 24 and 42 weeks
  Interventions: Device: NICAS cardiac output monitor
- Preterm infants: Preterm infants with fetal growth restriction
  Interventions: Device: NICAS cardiac output monitor

INTERVENTIONS:
Device: NICAS cardiac output monitor — Non-invasive continuous cardiac output monitoring device using total body bioimpedance.

SUMMARY:
This is an observational study in newborn term and preterm infants. The study will validate if non-invasive continuous cardiac output monitoring is feasible in newborn infants, if normative values can be constructed and what is the effect of fluid boluses and inotropes on cardiac output and peripheral vascular resistance.

DETAILED DESCRIPTION:
This is a 3-year prospective observational study.

Principal research question:

Is non-invasive continuous cardiac output (CO) measurement a validated tool of comprehensive cardiovascular assessment in neonatal intensive care (NICU)?

Secondary research questions:

1. Can robust normal ranges of CO be constructed for neonates undergoing cardiovascular measurement?
2. How do neonatal interventions (fluid boluses, ventilation and inotropes) affect CO?
3. Does the Non-invasive continuous cardiac output monitoring in children with foetal growth restriction (FGR) differ from normative CO data as above (1)?

A prospective study of stable newborn babies in the postnatal ward and sick term and preterm infants in the NICU in 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants in postnatal ward (within the first 72 hours of age)
* Term and Preterm infants (including those with FGR) admitted to the neonatal unit
* Written informed parental consent (prospective for postnatal ward and retrospective for babies admitted to the neonatal units)

Exclusion Criteria:

* Antenatal or postnatal diagnosis of severe congenital anomaly
* Infants with no realistic chance of survival
* Infants who are >12 hours of age
* Infants with fragile skin not permitting skin probe placement

Ages: 1 Hour to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All term and preterm infants (24-42 weeks of gestational age) for the validation study and preterm infants with fetal growth restriction for the longitudinal study.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Haemodynamic outcome comparison to echocardiography measured CO | 36 months
  Non-invasive continuous Cardiac Output (CO) measurement (mls/kg/min) during the first month of life in comparison to echocardiography measured CO (mls/kg/min)
Changes in cardiac output | 36 months
  Changes in cardiac output (CO) measurement (mls/kg/min) in relation to neonatal intervention

SECONDARY OUTCOMES:
Changes in clinical outcome - Survival at discharge | 36 months
  Survival at discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jayanta Banerjee, Principal Investigator — Neonatal consultant
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee J, Khatib N, Mansfield RC, Sathiyamurthy S, Kariholu U, Lees C. Continuous non-invasive measurement of cardiac output in neonatal intensive care using regional impedance cardiography: a prospective observational study. Arch Dis Child Fetal Neonatal Ed. 2024 Jun 19;109(4):450-455. doi: 10.1136/archdischild-2023-325941. PMID 38123965